CLINICAL TRIAL: NCT02936934
Title: Comparison of Adverse Drug Reactions Associated for Oxycodone and Morphine in Postoperative Pain After Abdominal Hysterectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital Civil de Guadalajara (Other)
Responsible Party: Principal Investigator, VIRGINIA ALEYDA SANCHEZ LOPEZ, MD Pharmacology, Hospital Civil de Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HospitalCG
Record Dates: First submitted 2016-10-14; First posted 2016-10-18 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-10

CONDITIONS: Pain, Postoperative
Keywords: Adverse Drug Reaction; Morphine; Oxycodone; Abdominal hysterectomy
MeSH Terms: conditions — Pain, Postoperative; Drug-Related Side Effects and Adverse Reactions | interventions — Morphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morphine (Active Comparator): Multimodal analgesia to morphine
  Interventions: Drug: Morphine
- Oxycodone (Experimental): Multimodal analgesia to oxycodone
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Morphine — Interventions pre-specified to be administered to participants:
  Abdominal hysterectomy Block Anesthesia: bupivacaine 0.5% + 25 micrograms of fentanyl 10mg / kg metamizol sodium intravenously during surgery
  Intravenous infusion:
  200μg / kg of morphine + 3g metamizole sodium + 3mg / kg 2% lidocaine + 500mL saline solution. Time administration:24hours
  Arms: Morphine
Drug: Oxycodone — Interventions pre-specified to be administered to participants:
  Abdominal hysterectomy Block Anesthesia: bupivacaine 0.5% + 25 micrograms of fentanyl 10mg / kg metamizol sodium intravenously during surgery
  Intravenous infusion:
  150μg / kg of oxycodone + 3g metamizole sodium + 3mg / kg 2% lidocaine + 500mL saline solution. Time administration: 24hours.
  Arms: Oxycodone

SUMMARY:
The objective of this study is compare adverse reactions associated with oxycodone and morphine for the treatment of postoperative pain after abdominal hysterectomy

DETAILED DESCRIPTION:
A randomized single-blind study, was performed to compare the adverse reactions associated with oxycodone and morphine in patients undergoing abdominal hysterectomy.

process:

1. A clinical history of patients candidates to participate in the study will be developed.
2. If you meet the selection criteria will be held the invitation to participate in the study, reading the letter under information

Patients who agree to participate in the study will be managet during the surgical procedure:

15 mg mixed blockade with bupivacaine 0.5% + 25 micrograms of fentanyl 10mg / kg intravenously during surgery metamizol 3) After the surgical procedure (immediate postoperative)

• the patient to group A or B (randomization) is assigned, masking infusions and allocation will be conducted by an outside person who will test an additional record the names of the patients and the drug administered.

A bolus of oxycodone or morphine 10% calculated dose for intravenous infusion 0.075mg intravenous palonosetron prophylaxis of emesis Detection and assessment of severity of adverse drug reactions will be conducted by an interview that will be at 0,1,2,6,12 and 24 hours after the onset of analgesia. Instrument designed for the detection of RAM will be used and classify its severity according to common terminology criteria for adverse events (CTCAE). Futhermore, measuring systemic blood pressure, heart rate, oxygen saturation will be performed through the use of Nihon Kohden monitor (model BSN-2301K). Pain assessment will be made by the numerical scale (NRS). The researcher responsible for the detection and assessment of adverse reactions to opioids and others determinations, remain mowed.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for abdominal hysterectomy
* Signing for informed consent

Exclusion Criteria:

* Patients used with MAO inhibitor drugs (<14 days before surgery)
* History of substance abuse
* Hypersensitivity to opioids and others drugs of multimodal analgesia (metamizol and lidocaine)
* Pretreatment of any opioid (<7/2 lives of the drug in question)
* Chronic pain of any etiology (> 6 months)
* Diagnosis of bowel obstruction
* Renal or hepatic insufficiency
* Asthma, chronic obstructive pulmonary disease (COPD), and/ or hypothyroidism.
* Patients requiring general anesthesia for surgical complications

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-02 (Estimated)

PRIMARY OUTCOMES:
Adverse drug reactions (questionnaire) | 24 hours
  Nausea, vomiting, respiratory depression, dizziness, headache, sedation, pruritus and anaphylaxis

SECONDARY OUTCOMES:
Postoperative pain (Numeric Pain Rating Scale) | 24 hours
systemic blood pressure (mmHg) (physiological parameter) | 24 hours
  Monitor Nihon Kohden BSM-2301K
Heart rate (physiological parameter) | 24 hours
  Monitor Nihon Kohden BSM-2301K
Oxygen saturation (physiological parameter) | 24 hours
  Monitor Nihon Kohden BSM-2301K

IPD SHARING:
Plan to Share IPD: No